CLINICAL TRIAL: NCT02840006
Title: Spinal Anesthesia Associated With General Anesthesia in Coronary Artery Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Gioielli de Castilho (Other)
Responsible Party: Sponsor-Investigator, Daniel Gioielli de Castilho, MD, Universidade do Vale do Sapucai
Organization: Universidade do Vale do Sapucai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MEDC
Record Dates: First submitted 2016-07-05; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Myocardial Revascularization; Spinal Anesthesia; Postoperative Care; Fentanyl
Keywords: Vasoconstrictor Agents; Vasodilator Agents
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anesthesia only (Active Comparator): Anesthetic induction with etomidate 0,3 a 0,4 mg.kg-1, citrate fentanyl 5 mcg.kg-1 and atracurium 0,5.kg-1
  Interventions: Procedure: General anesthesia only
- General anesthesia associated spinal anesthesia (Active Comparator): spinal anesthesia using bupivacaine 0,5% hyperbaric 20 mg, morphine 200 mcg, set trendeleburg for 10 minutes, sensitive test in T1. Anesthetic induction with etomidate 0,3 a 0,4 mg.kg-1, citrate fentanyl 5 mcg.kg-1 and atracurium 0,5.kg-1.
  Interventions: Procedure: General anesthesia and Spinal anesthesia

INTERVENTIONS:
Procedure: General anesthesia only — Induction drugs: Citrate of fentanyl, atracurium, etomidate
  Arms: General anesthesia only
Procedure: General anesthesia and Spinal anesthesia — Induction drugs: Citrate of fentanyl, atracurium, etomidate Spinal anesthesia: Bupivacaine hyperbaric, Morphine
  Arms: General anesthesia associated spinal anesthesia

SUMMARY:
CONTEXT: In patients eligible for coronary artery bypass surgery, anesthesia should provide a number of conditions that exceed the limits of cardiovascular stability, myocardial protection and other organs. Moreover, the combination of general anesthesia and spinal anesthesia lessens the homeostatic, metabolic, hormonal and immunosuppressive changes. The goal of this research was to evaluate the consumption of fentanyl citrate in intra-operative in Coronary Artery Bypass Grafting (CABG) surgery with cardiopulmonary bypass under spinal anesthesia associated with general anesthesia.

METHODS: Clinical, prospective, randomized and double covered study, approved by the Research Ethics Committee. Fifty-six patients candidates for CABG with CPB, after signing the Terms of consent, were randomized and divided into two groups: GI - General and GII - General + subarachnoid. General anesthesia was induced according to the weight of each patient and maintenance with isoflurane and fentanyl. Spinal anesthesia was induced with 20 mg of 0.5% hyperbaric bupivacaine and 200 mcg of morphine, the patient is placed in cephalo-position slope of 45 degrees for 10 minutes in Group II. In the statistical study was performed using the Mann-Whitney test; the level of statistical significance was set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* Underwent cardiac artery bypass surgery with cardiopulmonary bypass, with
* No restriction on age
* No restriction on ethnicity
* No restriction on education or social class

Exclusion Criteria:

* Patients with sternotomy provided; those
* Urgent surgery and/or emergency
* Patient was with signs of shock
* Patients with chronic renal failure
* Patients with liver disorders
* Tracheostomy patients
* Patients with presence of use of mechanical ventilatory support;
* Patients with physical disabilities; bedridden and wheelchair users.
* Patients to withdraw the Consent and Informed
* Patients who eventually had to be re-operated in the presence also of the mechanical ventilatory support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
consumption of fentanyl citrate in intra-operative in Coronary Artery Bypass Grafting surgery with cardiopulmonary bypass under spinal anesthesia associated with general anesthesia. | in 24 hours
  Will be measure the consumption of fentanyl in 24 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital das Clinicas Samuel Libânio, Pouso Alegre, Minas Gerais
  - Univas, Pouso Alegre, Minas Gerais

IPD SHARING:
Plan to Share IPD: Yes